CLINICAL TRIAL: NCT02676141
Title: Responsiveness of the German Version of the Neck Disability Index (NDI-G)
Status: Completed | Type: Observational
Sponsor: Balgrist University Hospital (Other)
Collaborators: Maastricht University (Other)
Responsible Party: Principal Investigator, Swanenburg, Head of PT Research, Balgrist University Hospital
Other Study IDs: 2015-00068
Record Dates: First submitted 2016-01-29; First posted 2016-02-08 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Neck Pain Chronic
MeSH Terms: interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Manual Therapy — The treatment the patients receive is not specifically set up for the study. Participants will already be seeing a practitioner before the participants are included in the study.

SUMMARY:
This study evaluates if the German Version of the NDI is sensitive to change over time.

DETAILED DESCRIPTION:
Chronic neck pain patients will be asked to participate in the study.

The participants are asked to fill out the NDI at the beginning of the study and after seven weeks. Additionally the participants will fill out the PGIC.

ELIGIBILITY:
Inclusion Criteria:

* Chronic neck pain
* over 18 years old
* informed consent
* able to speak, write and read German.

Exclusion Criteria:

* Any problems that may exclude Manual Therapy treatment of the cervical spine e.g fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic neck pain.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-02-10 (Actual)

PRIMARY OUTCOMES:
Change of the German Version of the Neck Disability Index (NDI-G) | Change from Baseline to seven weeks
  Questionnaire to evaluate the subjective restriction of the participants

SECONDARY OUTCOMES:
Patient's Global Impression of Change Scale (PGIC) | Seven weeks after the baseline measurement
  Questionnaire measuring the change of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Jaap Swanenburg, PhD, Principal Investigator — Balgrist University Hospital
Locations (1):
- Balgrist University Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Langenfeld A, Gassner AP, Wirth B, Muhlemann MB, Nyiro L, Bastiaenen C, Swanenburg J. Responsiveness of the German version of the Neck Disability Index in chronic neck pain patients: a prospective cohort study with a seven-week follow-up. Arch Physiother. 2022 Oct 17;12(1):23. doi: 10.1186/s40945-022-00149-y. PMID 36244985